CLINICAL TRIAL: NCT04126707
Title: A Single-center, Open-label, Single-dose Phase I Study to Investigate the Absorption, Metabolism and Excretion of [14C] HQP1351 After a Single Oral 30mg (100µCi) Dose in Healthy Chinese Male Subjects
Brief Title: The Absorption, Metabolism and Excretion of [14C] HQP1351 in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: HealthQuest Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQP1351XC105
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2020-07

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: Chronic Myeloid Leukemia; HQP1351
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] HQP1351 (Experimental): To investigate the absorption properties, as well as to evaluate the mass balance and elucidate the pathways of biotransformation after a single oral dose (30mg, 100µCi) of [14C] HQP1351 to healthy Chinese male subjects.
  Interventions: Drug: [14C] HQP1351

INTERVENTIONS:
Drug: [14C] HQP1351 — Orally, single dose of 30mg

SUMMARY:
The objective of this study is to determine the mass balance and routes of excretion of total radioactivity after a single oral 30mg (100µCi) dose of [14C] HQP1351 given as a suspension. For further clinical development, human mass balance data are required to elucidate the absorption, metabolism, and excretion of HQP1351.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if he meets the following criteria:

1. Healthy male volunteers between the ages of 18 to 50 years old, inclusive;
2. Body weight >=50 kg, Body mass index (body weight(kg)/hight2(m2)) between 19 and 26 kg/m2 (inclusive);
3. Normal physical findings, clinical laboratory values, vital signs and 12-lead ECG, or any abnormality that is non-clinically significant;
4. Male subjects of reproductive potential with partners will be instructed to, and must be willing to practice a highly effective method of birth control for the duration of the study and continuing 1 year after discontinuing treatment with the investigational product.
5. Must understand, and voluntarily sign the informed consent, comply with the requirements of the study.

Exclusion Criteria:

A subject will not be eligible for study participation if he meets any of the exclusion criteria:

1. History of or current clinically significant cardio, pulmonary, endocrine, metabolism, renal, hepatic, gastrointestinal, dermatology, infection, hematology, neurological, mental disease or disorder;
2. Positive test for HBsAg, HBeAg, anti-HCV, anti-HIV or syphilis antibody;
3. Abnormality in blood pressure, including hypertensive BP (SBP>=140 mmHg, or DBP >=90 mmHg), or hypotensive BP (SBP<90 mmHg, or DBP <=55 mmHg), Pulse rate<55 bpm or >100 bpm;
4. Long-QT syndrome or family history of it, or QTcB interval > 450 ms; intraventricular blocks or left/right bundle branch block or QRS>120ms; frequent ventricular ectopic beats (any 10s ECG ventricular premature beat >= 1 in screening period); or abnormal resting heart rate (> 100 bpm)
5. The following abnormal clinical laboratory values

   1. HGB < LLN or HGB>ULN, and is judged as clinically significant by the investigator；
   2. Abnormal ALB, TP, CRE, ALT, AST, BIL, BUN, GLU value, and is judged as clinically significant by the investigator;
6. Received any drug within 14 days before taking the investigational drug, including any prescription drug, OTC drug, herbal drug or health care product with medicinal effect;
7. Received any other investigating products or participated in any clinical trails three month before screening or within 10 t1/2 after receiving other investigating products;
8. History of or current swallowing disorder, active gastrointestinal diseases, or other diseases that significantly affect absorption, distribution, metabolism and excretion of drugs;
9. Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease or history of gastrointestinal surgery and cholecystectomy;
10. Hemorrhoids or perianal disease with regular/perianal bleeding;
11. Allergies, have allergies to two or more drugs or foods; or have known allergies to the components of the drug (microcrystalline cellulose, stearic acid, croscarmellose sodium);
12. Have donated 400ml or more of blood or plasma 3 months prior to the study drug administration, or more than 50ml within 2 weeks prior to administration;
13. Vaccination was administered within 6 months prior to screening or during screening;
14. History of drug or alcohol abuse;
15. Smoking (> 10 cigarette / day), drinking (> 15 g, pure alcohol / day, equivalent to 450 ml beer, 150 ml wine or 50 ml low-alcohol liquor), or abusing drugs within last 3 months;
16. Subject with mentally ill and could not understand the property, scope and possible consequences of the study;
17. subject in prison or whose freedom is restricted by administrative or legal issues;
18. Failure to comply with clinical study protocols, such as non-cooperation, follow-up visit and completion of entire study;
19. Abnormal coagulation function or known severe bleeding tendency;
20. Subjects who have participated in radiolabeled clinical study prior to drug administration;
21. Significant radiation exposure within one year prior to drug administration (more than one exposure from chest X-ray, CT scan, or barium meal examination and radiation-related occupations).
22. Investigators think that subjects are not suitable to participate in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 6 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Radioactivity concentration of each blood and plasma sample | Day 1- Day 15
  Use liquid scintillation counter to evaluate Radioactivity concentration of each blood and plasma sample
Radioactivity concentration of each urine samples | Day 1- Day 15
  Use liquid scintillation counter to evaluate Radioactivity concentration of each urine sample
Radioactivity concentration of each feces samples | Day 1- Day 15
  Use liquid scintillation counter to evaluate Radioactivity concentration of each feces sample
Total recovery of radioactivity in urine and feces | Day 1- Day 15
  Calculate the total radioactivity in urine and feces based on the radioactivity concentration of each sample

SECONDARY OUTCOMES:
Plasma drug concentrations | Day 1- Day 15
  To determine the plasma concentrations of HQP1351 with validated LC-MS/MS method for obtaining its pharmacokinetics parameters
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Day 1- Day 15
  According to CTCAE v5.0, the number and frequency of adverse events after a single dose of test drug were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shao, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, China